CLINICAL TRIAL: NCT03931616
Title: Berlin PRehospital Or Usual Delivery of Acute Stroke Care 2.0
Brief Title: Berlin PRehospital Or Usual Delivery of Acute Stroke Care 2.0 (B_PROUD 2.0)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Center for Stroke Research Berlin (Other)
Responsible Party: Principal Investigator, Heinrich J Audebert, Prof. Dr. med., MD, Neurologist, Head of Dept. of Neurology at Campus Benjamin Franklin, Charité - Universitaetsmedizin Berlin, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B_PROUD 2.0
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Stroke
Keywords: stroke; prehospital; telemedicine; thrombolysis; endovascular treatment; functional outcome
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEMO deployment (Experimental): STEMOs are specialized stroke ambulances providing prehospital neurovascular expertise, a CT scanner, point-of-care testing, and telemedical support.
  Interventions: Procedure: STEMO
- Regular care (Active Comparator): Regular prehospital care consists of normal ambulance care. In suspected life-threatening cases, an emergency physician is sent to the emergency scene in parallel.
  Interventions: Procedure: Regular care

INTERVENTIONS:
Procedure: STEMO — STEMO, the intervention, includes prehospital neurological emergency assessment with the option to perform CT and CT-angiography, start specialized treatment at the door-step of the patient's house, including thrombolysis with tissue Plasminogen Activator and blood pressure management (choice of drug at discretion of treating physician), use of telemedicine for image transfer as well as results of point-of-care laboratory, prenotification (e.g. for endovascular treatment), triage and transport.
  Arms: STEMO deployment
Procedure: Regular care — A regular ambulance, the comparator, not equipped with advanced point-of-care laboratory or CT scanner, without telemedicine and not staffed with a neurologist.
  Arms: Regular care

SUMMARY:
Prehospital stroke care in specialized ambulances increases thrombolysis rates, reduces alarm-to-treatment times, and improves prehospital triage. Preliminary analyses suggest cost-effectiveness. However, scientific proof of improved functional outcome compared to usual care is still lacking. The objective of this trial is to show improved functional outcomes after deployment of a Stroke Emergency Mobile (STEMO) compared to regular care.

DETAILED DESCRIPTION:
This is a pragmatic, prospective, multi-center trial with blinded outcome assessment of treatment candidates three months after stroke. Treatment candidates will be defined as patients with final discharge diagnosis of cerebral ischemia, and onset-to-alarm time ≤4 hours, disabling symptoms not resolved at time of ambulance arrival, and able to walk without assistance prior to emergency. These patients will be included if their emergency call from a predefined catchment area in Berlin, Germany, caused a stroke alarm at the dispatch center during STEMO hours (7am-11pm, Monday-Sunday). About 50% of STEMO dispatches will be handled by regular ambulances since STEMO will be already in operation creating the quasi-randomized control group.

Because of several organisational issues during the transition of the STEMO service into provisional regular care, the B_PROUD 1.0 evaluation has been defined as implementation study and will be complemented by the B_PROUD 2.0 study. B_PROUD 2.0. recruits patients with index event after May 1st, 2019.

B_PROUD uses data from the Berlin - SPecific Acute Treatment in ischemic and hemorrhagIc Stroke with longterm outcome (B-SPATIAL) registry. The B-SPATIAL registry started recruitment in January 2016.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected acute stroke according to the dispatcher stroke identification algorithm during STEMO hours (7am-11pm, Monday-Sunday) and within the STEMO catchment area

   Inclusion criteria for primary study population:
2. Final diagnosis of ischemic stroke (ICD 10: I63) or TIA (Transient Ischemic Attack, ICD 10: G45 except G45.4)
3. Confirmed onset-to-alarm time ≤ 4 hours at dispatch
4. Pre-stroke modified Rankin scale ≤ 3 (being able to ambulate, in routine clinical care, patients with mRS up to 3 are usually deemed suitable for tissue plasminogen activator treatment)

Exclusion Criteria:

1. Remission of disabling symptoms until arrival of emergency medical service
2. Malignant or other severe primary disease with life expectancy < 1 year

   Additional exclusion criteria for primary study population:
3. Major surgery within 4 weeks before study inclusion
4. Confirmed stroke within 3 months before study inclusion
5. Absolute contraindications for thrombolysis AND thrombectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale | 3 months
  Assessment of functional outcome over the entire range of the modified Rankin Scale. The scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Co-primary 3-Month Outcome | 3 months
  The co-primary 3-month outcome includes the following range of outcomes:
  1. mRS 1-3 if available or living at home (information according registration office at 4 month after stroke)
  2. mRS 4-5 or (if mRS is missing) living in institution (information according registration office at 4 month after stroke)
  3. death.
  The co-primary outcome will only be used if the mRS follow-up rate remains below 91%. This will help to include valuable information for patients without concrete mRS follow-up information. All outcomes will be calculated with ordinal logistic regression.

SECONDARY OUTCOMES:
Thrombolysis rate | 3 months
Thrombectomy rate | 3 months
Diagnosis and treatment times (D) | 3 months
  alarm-to-treatment time
Diagnosis and treatment times (A) | 3 months
  Onset-to-treatment time
Diagnosis and treatment times (B) | 3 months
  onset-to-reperfusion time (for thrombectomy)
Diagnosis and treatment times (C) | 3 months
  alarm-to-imaging time
Diagnosis and treatment times (E) | 3 months
  imaging-to-treatment time
Cost-effectiveness (A) | 3 months
  Additional costs due to implementation and running of STEMO
Cost-effectiveness (B) | 3 months
  duration of hospital stay regarding acute treatment and rehabilitation
Cost-effectiveness (C) | 3 months
  hospital related costs
Cost-effectiveness (D) | 3 months
  costs of long-term care based on projections
Cost-effectiveness (E) | 3 months
  Additional costs due to implementation and running of STEMO, duration of hospital stay regarding acute treatment and rehabilitation, hospital related costs, costs of long-term care based on projections
Quality of life | 3 months
  Assessment with European Quality of Life - 5 Dimensions (EQ-5D)
Modified Rankin Scale shift analyses | 3 months
  Shift analyses for mRS ≤ 1 at 3 months in patients ≤ 80 years of age living at home without disability and mRS ≤ 2 at 3 months in patients > 80 years of age or living at home with help or living in an Institution.
  For a detailed description of the modified Rankin Scale (mRS) see 1.
In-hospital mortality | 7 days
  Frequency of patients dying within the duration of the hospital stay after admission for stroke.
Death rate over time | 3 months
  Deaths over time will be determined and compared between groups using a Kaplan-Meier plot
Discharge status | 3 months
  Including in-hospital mortality among patients not included in the primary study population (patients with intracranial hemorrhages as well as patients receiving thrombolysis in stroke mimics)
Modified Rankin Scale in patients with intracranial hemorrhages | 3 months
  Assessment of functional outcome among patients with intracranial hemorrhages.
  For a detailed description of the modified Rankin Scale (mRS) see 1.
Rate of secondary emergency medical service deliveries to specialized facilities | 3 months
  Assessment for patients with acute ischemic stroke to hospitals with Stroke Unit, for patients with cerebral artery occlusion (internal carotid artery, M1 or proximal M2 segment of middle cerebral artery) to hospitals with thrombectomy facility, and for patients with intracerebral hemorrhage to hospitals with neurosurgery department.
Symptomatic hemorrhage (A) | 3 months
  According to clinical categorisation as documented in discharge letters within 36 hours of treatment in patients receiving thrombolysis or thrombectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Charité, Berlin, Germany

REFERENCES:
- [Background] Ebinger M, Winter B, Wendt M, Weber JE, Waldschmidt C, Rozanski M, Kunz A, Koch P, Kellner PA, Gierhake D, Villringer K, Fiebach JB, Grittner U, Hartmann A, Mackert BM, Endres M, Audebert HJ; STEMO Consortium. Effect of the use of ambulance-based thrombolysis on time to thrombolysis in acute ischemic stroke: a randomized clinical trial. JAMA. 2014 Apr 23-30;311(16):1622-31. doi: 10.1001/jama.2014.2850. PMID 24756512
- [Background] Krebes S, Ebinger M, Baumann AM, Kellner PA, Rozanski M, Doepp F, Sobesky J, Gensecke T, Leidel BA, Malzahn U, Wellwood I, Heuschmann PU, Audebert HJ. Development and validation of a dispatcher identification algorithm for stroke emergencies. Stroke. 2012 Mar;43(3):776-81. doi: 10.1161/STROKEAHA.111.634980. Epub 2012 Jan 5. PMID 22223240
- [Background] Ebinger M, Fiebach JB, Audebert HJ. Mobile computed tomography: prehospital diagnosis and treatment of stroke. Curr Opin Neurol. 2015 Feb;28(1):4-9. doi: 10.1097/WCO.0000000000000165. PMID 25490196
- [Background] Wendt M, Ebinger M, Kunz A, Rozanski M, Waldschmidt C, Weber JE, Winter B, Koch PM, Freitag E, Reich J, Schremmer D, Audebert HJ; STEMO Consortium. Improved prehospital triage of patients with stroke in a specialized stroke ambulance: results of the pre-hospital acute neurological therapy and optimization of medical care in stroke study. Stroke. 2015 Mar;46(3):740-5. doi: 10.1161/STROKEAHA.114.008159. Epub 2015 Jan 29. PMID 25634000
- [Background] Kunz A, Ebinger M, Geisler F, Rozanski M, Waldschmidt C, Weber JE, Wendt M, Winter B, Zieschang K, Fiebach JB, Villringer K, Erdur H, Scheitz JF, Tutuncu S, Bollweg K, Grittner U, Kaczmarek S, Endres M, Nolte CH, Audebert HJ. Functional outcomes of pre-hospital thrombolysis in a mobile stroke treatment unit compared with conventional care: an observational registry study. Lancet Neurol. 2016 Sep;15(10):1035-43. doi: 10.1016/S1474-4422(16)30129-6. Epub 2016 Jul 16. PMID 27430529
- [Background] Ebinger M, Harmel P, Nolte CH, Grittner U, Siegerink B, Audebert HJ. Berlin prehospital or usual delivery of acute stroke care - Study protocol. Int J Stroke. 2017 Aug;12(6):653-658. doi: 10.1177/1747493017700152. Epub 2017 Mar 22. PMID 28649936
- [Background] Kunz A, Nolte CH, Erdur H, Fiebach JB, Geisler F, Rozanski M, Scheitz JF, Villringer K, Waldschmidt C, Weber JE, Wendt M, Winter B, Zieschang K, Grittner U, Kaczmarek S, Endres M, Ebinger M, Audebert HJ. Effects of Ultraearly Intravenous Thrombolysis on Outcomes in Ischemic Stroke: The STEMO (Stroke Emergency Mobile) Group. Circulation. 2017 May 2;135(18):1765-1767. doi: 10.1161/CIRCULATIONAHA.117.027693. No abstract available. PMID 28461420
- [Derived] Rohmann JL, Piccininni M, Ebinger M, Wendt M, Weber JE, Schwabauer E, Freitag E, Zuber M, Bernhardt L, Lange J, Erdur H, Behrens J, Ganeshan R, Schlemm L, Harmel P, Liman TG, Lorenz-Meyer I, Rohrpasser-Napierkowski I, Hille A, Bohner G, Nabavi DG, Schmehl I, Ekkernkamp A, Jungehulsing GJ, Mackert BM, Hartmann A, Endres M, Audebert HJ. Effect of Mobile Stroke Unit Dispatch on Process Parameters and Functional Outcomes in Patients With Acute Stroke: The B_PROUD-2.0 Study. Neurology. 2025 Nov 11;105(9):e214225. doi: 10.1212/WNL.0000000000214225. Epub 2025 Oct 16. PMID 41100781
- [Derived] Harmel P, Ebinger M, Freitag E, Grittner U, Lorenz-Meyer I, Napierkowski I, Nolte CH, Siegerink B, Audebert HJ. Functional stroke outcomes after mobile stroke unit deployment - the revised protocol for the Berlin Prehospital Or Usual Delivery of acute stroke care (B_PROUD) part 2 study. Neurol Res Pract. 2019 Jun 3;1:18. doi: 10.1186/s42466-019-0022-4. eCollection 2019. PMID 33324884
- See also: Prehospital Thrombolysis: A Manual from Berlin (2013) — http://www.jove.com/video/50534/prehospital-thrombolysis-a-manual-from-berlin